CLINICAL TRIAL: NCT02223572
Title: Secondary Fracture Prevention in Patients Hospitalized for Hip Fracture: Adding the Metabolic Treatment to the Surgical One.
Brief Title: Secondary Fracture Prevention in Patients Who Suffered From Osteoporotic Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: pninarotman (Other)
Collaborators: Meir Medical Center (Other)
Responsible Party: Sponsor-Investigator, pninarotman, Depart. of Medicine 'E' Deputy Head, Meir Medical Center
Organization: Meir Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HipFracture2014
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Hip Fractures; Osteoporotic Fractures; Osteoporosis
MeSH Terms: conditions — Hip Fractures; Osteoporotic Fractures; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- osteoporotic hip fracture (Experimental)
  Interventions: Radiation: hip Xray

INTERVENTIONS:
Radiation: hip Xray

SUMMARY:
Due to its prevalence worldwide, osteoporosis is considered a serious public health concern. The worldwide annual incidence of Osteoporotic fractures is approximately 2 million in the US only.

Hip fracture is associated with serious disability and excess mortality. Studies have shown that an initial osteoporotic fracture is a major risk factor for a new fracture. An increased risk of 14.8% for a secondary hip fracture has been demonstrated in people that have already sustained a fracture in the past 4 years (In average). These data indicate the major opportunity afforded by secondary fracture prevention strategies.

By responding to the first fracture, we can reduce the incidence of second and subsequent fractures. However, even after longer medical follow-up according to regular standard of care, medical treatment and rehabilitation, the medical system has been unable to translate the eminent risk into an effective preventive treatment.

DETAILED DESCRIPTION:
Study Objectives:

* To create a treatment, follow up and rehabilitation protocol for patients who suffered from a hip fracture, in order to prevent a secondary fracture.
* To demonstrate that a combined treatment from the Hip Fractures Clinic as well as the regular standard treatment and rehabilitation suggested by the Bone Health Clinic (both in addition to standard medication prescribed for osteoporosis) will result in a significant reduction of second and subsequent fractures.

Study Protocol:

1. The study protocol will begin after the patients, who have been admitted with a primary hip fracture (of osteoporotic nature), were surgically treated (as customary standard of care).
2. According to hospitalization standard protocol, the patients will be treated with vitamin D and calcium. For the first month the patient will be given a loading dose of 70,000 units. For the next months the patients will receive 50,000-80,000 units per month.

   In addition, the patient will be treated with Calcium Pills (Caltrate TAB 600mg, once a day)
3. In addition to the clinical customary monitoring tests performed during the hospitalization, Biomarkers and safety assessment will be taken:

   1. Vitamin D
   2. Bone Markers - Bone markers will be taken three days after the patient was admitted, and one more time six months later (as part of follow up visit).
4. Follow up visits after hospitalization due to surgery for primary hip fracture.

   1. Follow up visits at the Hip Fracture Clinic will occur in intervals of: six weeks, 3 months, 6 months and a year, since the patient had been released from hospitalization. At follow up visit, the patient will be assessed for physical examination, hip X-ray and the rehabilitation progression Questionnaire (HHS).
   2. Follow up visits at the Bone Health Clinic will occur between 6 weeks to 3 months since the patient had been released from hospitalization (as part of regular standard of care).
   3. A 3cc Serum sample will be taken with the purpose to serve on future studies and examine new markers such as bone markers SCLEROSTIN. There will be no further use of these samples. The samples will remain in deep freeze temperature (C˚70-).

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years old
* Patients diagnosed with low energy osteoporotic hip fracture, and was treated under surgery.

Exclusion Criteria:

* Patients not diagnosed with osteoporosis.
* Patients diagnosed with high energy osteoporotic hip fracture.
* Patients that suffered from Multiple Trauma.
* Patients diagnosed with Metabolic diseases or Genetic diseases.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Reduce number of incidents of secondary hip fracture. | 1 year and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Yaacobi, M.D., Principal Investigator — Meir Medical Center; Pnina Rotman, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel, Israel